CLINICAL TRIAL: NCT04043104
Title: A Phase 1 Open-Label, Dose Escalation Study to Determine the Optimal Dose, Safety, and Activity of AAV2hAQP1 in Subjects With Radiation-Induced Parotid Gland Hypofunction and Xerostomia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MeiraGTx UK II Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MGT016
Record Dates: First submitted 2019-07-23; First posted 2019-08-02 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Radiation-Induced Parotid Gland Hypofunction; Xerostomia Due to Radiotherapy; Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- 1 x 10^11 vg/gland (single gland) (Experimental)
  Interventions: Drug: AAV2hAQP1: 1 x 10^11 vg/gland (single gland)
- 3 x 10^10 vg/gland (both glands) (Experimental)
  Interventions: Drug: AAV2hAQP1: 3 x 10^10 vg/gland (both glands)
- 3 x 10^11 vg/gland (single gland) (Experimental)
  Interventions: Drug: AAV2hAQP1: 3 x 10^11 vg/gland (single gland)
- 1 x 10^11 vg/gland (both glands) (Experimental)
  Interventions: Drug: AAV2hAQP1: 1 x 10^11 vg/gland (both glands)
- 1 x 10^12 vg/gland (single gland) (Experimental)
  Interventions: Drug: AAV2hAQP1: 1 x 10^12 vg/gland (single gland)
- 3 x 10^11 vg/gland (both glands) (Experimental)
  Interventions: Drug: AAV2hAQP1: 3 x 10^11 vg/gland (both glands)
- 3 x 10^12 vg/gland (single gland) (Experimental)
  Interventions: Drug: AAV2hAQP1: 3 x 10^12 vg/gland (single gland)
- 1 x 10^12 vg/gland (both glands) (Experimental)
  Interventions: Drug: AAV2hAQP1: 1 x 10^12 vg/gland (both glands)

INTERVENTIONS:
Drug: AAV2hAQP1: 1 x 10^11 vg/gland (single gland) — Intra-parotid administration of AAV2hAQP1 via Stensen's duct to a single parotid gland at a dose level of 1 x 10^11 vg/gland
  Arms: 1 x 10^11 vg/gland (single gland)
Drug: AAV2hAQP1: 3 x 10^10 vg/gland (both glands) — Intra-parotid administration of AAV2hAQP1 via Stensen's duct to both parotid glands at a dose level of 3 x 10^10 vg/gland
  Arms: 3 x 10^10 vg/gland (both glands)
Drug: AAV2hAQP1: 3 x 10^11 vg/gland (single gland) — Intra-parotid administration of AAV2hAQP1 of via Stensen's duct to a single parotid gland at a dose level of 3 x 10^11 vg/gland
  Arms: 3 x 10^11 vg/gland (single gland)
Drug: AAV2hAQP1: 1 x 10^11 vg/gland (both glands) — intra-parotid administration of AAV2hAQP1 via Stensen's duct to both parotid glands at a dose level of 1 x 10^11 vg/gland
  Arms: 1 x 10^11 vg/gland (both glands)
Drug: AAV2hAQP1: 1 x 10^12 vg/gland (single gland) — Intra-parotid administration of AAV2hAQP1 via Stensen's duct to a single parotid gland at a dose level of 1 x 10^12 vg/gland
  Arms: 1 x 10^12 vg/gland (single gland)
Drug: AAV2hAQP1: 3 x 10^11 vg/gland (both glands) — Intra-parotid administration of AAV2hAQP1 via Stensen's duct to both parotid glands at a dose level of 3 x 10^11 vg/gland
  Arms: 3 x 10^11 vg/gland (both glands)
Drug: AAV2hAQP1: 3 x 10^12 vg/gland (single gland) — Intra-parotid administration of AAV2hAQP1 via Stensen's duct to a single parotid gland at a dose level of 3 x 10^12 vg/gland
  Arms: 3 x 10^12 vg/gland (single gland)
Drug: AAV2hAQP1: 1 x 10^12 vg/gland (both glands) — Intra-parotid administration of AAV2hAQP1 via Stensen's duct to both parotid glands at a dose level of 1 x 10^12 vg/gland
  Arms: 1 x 10^12 vg/gland (both glands)

SUMMARY:
Open-label, non-randomized, dose escalation trial of AAV2hAQP1 administered via Stensen's duct to a single or both parotid glands in subjects with radiation-induced xerostomia The objectives are to evaluate the safety and identify either a maximum tolerated dose or a maximum feasible dose of a single dose of AAV2hAQP1 infused into one or both parotid glands:

To evaluate subject improvement of xerostomia symptoms, to evaluate the increase in parotid gland salivary output after treatment with AAV2hAQP1, to evaluate additional efficacy outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥18 years of age.
2. History of radiation therapy for head and neck cancer.
3. Abnormal parotid gland function as judged by both absence of unstimulated parotid salivary flow and a stimulated parotid salivary flow in the targeted parotid gland >0 and <0.3 mL/min/gland after 2% citrate stimulation.
4. No evidence of recurrence of the primary malignancy by an otolaryngology (ears, nose, and throat [ENT]) assessment. Additionally, all subjects must be disease-free of head and neck cancer for at least 5 years following the end of treatment at screening, with the exception of subjects with a history of HPV+ OPC (base of tongue, oropharynx, pharynx, soft palate, tonsil) who must be disease free for at least 2 years following the end of treatment. Disease status will be determined by negative clinical examinations and computed tomography (CT) scans of the neck and chest. If subjects have had a magnetic resonance imaging (MRI) of the neck or a positron emission tomography (PET) scan within 6 months of screening, then a CT scan is not required, except for HPV+ OPC subjects who must have scans at 2 years post treatment.
5. Female subjects of childbearing potential (i.e., ovulating, pre-menopausal, and not surgically sterile) and all male subjects must use a medically accepted contraceptive regimen during their participation in the study and until all samples collected at 2 consecutive visits following AAV2hAQP1 administration are negative. Acceptable methods of contraception for male subjects include the following:

   * Condoms with spermicide. Acceptable methods of contraception for female subjects include the following:
   * Intrauterine device for at least 12 weeks prior to Screening.
   * Hormonal contraception (oral, implant, injection, ring, or patch) for at least 12 weeks prior to Screening.
   * Diaphragm used in combination with spermicide.

Exclusion Criteria:

1. Pregnant or lactating women or women planning to become pregnant.
2. Any experimental therapy within 3 months before Day 1.
3. Active infection that requires the use of intravenous antibiotics and does not resolve at least 1 week before Day 1.
4. Uncontrolled ischemic heart disease (i.e., unstable angina, evidence of active ischemic heart disease on electrocardiogram [ECG]).
5. History of systemic autoimmune diseases affecting the salivary glands.
6. Use of systemic immunosuppressive medications (i.e., corticosteroids).

   o Note: Topical, inhaled, or intranasal corticosteroids are allowed.
7. Malignancy, other than head and neck cancer, within the past 3 years, with the exception of adequately treated basal cell or squamous cell carcinoma of the skin or in situ cervical carcinoma.
8. Active infections including, Epstein-Barr virus (EBV), cytomegalovirus (CMV), hepatitis B (HBV), hepatitis C (HCV), or human immunodeficiency virus (HIV) infection.
9. White blood cell count <3000/μL, absolute neutrophil count <1500/μL, hemoglobin <10.0 g/dL, platelet count <100,000/μL, or absolute lymphocyte count ≤500/μL.
10. Alanine aminotransferase and/or aspartate aminotransferase >1.5 × the upper limit of normal (ULN), alkaline phosphatase >1.5 × ULN, or total bilirubin >1.5 × ULN with any elevation of liver enzymes.
11. Estimated glomerular filtration rate <60 mL/min/1.73 m2 using the Modification of Diet in Renal Disease equation.
12. Active use of tobacco products as determined by self-reporting.
13. Allergy to iodine or shellfish, and thus unable to have sialographic evaluations.
14. Allergy or hypersensitivity to glycopyrrolate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-06-30 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
The primary outcome is safety of AAV2hAQP1 administered to the parotid gland of adult subjects with radiation-induced xerostomia | one day to one year
  Safety will be assessed by number of adverse events occurring with treatment

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - Leland Stanford Junior University, Stanford, California
  - University of Louisville, Louisville, Kentucky
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Atrium Health, Charlotte, North Carolina
- Health Sciences North - Northeast Cancer Center, Greater Sudbury, Ontario, Canada